CLINICAL TRIAL: NCT06113952
Title: A MULTICENTER LOW-INTERVENTIONAL STUDY TO EVALUATE AND MONITOR TREATMENT EXPERIENCE WITH WEEKLY GROWTH HORMONE (NGENLA) VERSUS DAILY GROWTH HORMONE INJECTIONS IN CHILDREN WITH GROWTH HORMONE DEFICIENCY
Brief Title: A Study to Compare the Experiences of Taking Daily Growth Hormone Injections to Weekly Ngenla in Children With Low Levels of Growth Hormone
Status: Withdrawn | Type: Observational
Why Stopped: company business-strategic decision
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C0311024
Record Dates: First submitted 2023-10-05; First posted 2023-11-02 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-10

CONDITIONS: Pediatric Growth Hormone Deficiency
Keywords: adherence; pediatric; Ngenla; growth hormone; growth hormone deficiency; daily growth hormone; smart bin; treatment experience
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with weekly growth hormone: Approximately 200 children with a diagnosis of pGHD who are treatment naïve or currently receiving once weekly Ngenla will be enrolled.
  Interventions: Device: Sharps bin to collect used needles/injections
- Patients treated with daily growth hormone: Approximately 200 children with a diagnosis of pGHD who are treatment naive or currently receiving daily GH injections will be enrolled
  Interventions: Device: Sharps bin to collect used needles/injections

INTERVENTIONS:
Device: Sharps bin to collect used needles/injections — Enrolled participants will be provided with a Smart Sharps Bin. The bin will collect used needles over a period of 12 months starting from enrollment.

SUMMARY:
The purpose of this study is to learn about:

* how children stick to taking their injections
* their experience with the study medicines (Ngenla and daily growth hormone) prescribed to children with low levels of growth hormone.

This study is seeking participants who:

* are being treated or are ready to start treatment with daily growth hormone or Ngenla.
* use a sharps bin to collect used needles.

The study medicines will be given as per regular care agreed with the doctor. The study will compare participant experiences to help us see:

- the difference in how the participants stick to taking their daily growth hormone injections compared to participants using once weekly Ngenla.

Participants will take part in this study for up to 14 months. During this time, they will have 3 study visits at the study clinic. The participants will use the HealthBeacon™ smart sharps bin for collecting the used needles or injections.

DETAILED DESCRIPTION:
This multicenter, international, longitudinal, prospective, site-based, low-interventional study aims to evaluate and monitor treatment experience, defined by treatment adherence and persistence, in children aged 3-16 years old with a diagnosis of pediatric growth hormone deficiency (pGHD), receiving either daily growth hormone (dGH) treatment or once weekly Ngenla. The study is planned to be conducted in a total of 50 participating sites distributed across Belgium, Canada, France, Italy, Luxembourg, Spain, UK, and US.

Data on treatment adherence and persistence will be collected in real-time over a period of 12 months using the HealthBeacon™ Smart Sharps Bin™ as a treatment monitoring device.

Additional data, including demographic and clinical characteristics, will be collected at three timepoints, in line with the routine care in each participating site and/or country, over a maximum period of 14 months.

Approximately 400 participants will be enrolled in the study (approximately 200 participants prescribed dGH injections and approximately 200 prescribed Ngenla).

ELIGIBILITY:
Inclusion Criteria:

1. Children of any sex aged 3-16 years at baseline
2. Children that have received a diagnosis of pGHD requiring GH injections.
3. Children that are currently being treated (dGH/Ngenla) or are treatment naïve but ready to start treatment.
4. Those who currently use a sharps bin to collect used needles [as per normal standard of care (SoC)].

Exclusion Criteria:

1. Children with psychosocial dwarfism.
2. Children born small for gestational age (SGA)
3. Children with chromosomal abnormalities
4. Children with other causes of short stature, such as uncontrolled primary hypothyroidism or rickets.
5. Children with a history of cancer.

7. Children with other acute medical or psychiatric condition

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients diagnosed with pGHD who are currently receiving growth hormone treatment or are about to start it.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-10-17 (Estimated); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Mean Adherence To Ngenla and daily growth hormone | 12 months
  The adherence for Ngenla and daily growth hormone followed the medication possession ratio definition(MPR). The MPR is calculated from the total number of injections used and collected in the Smart Sharps Bin™ .

SECONDARY OUTCOMES:
Percentage of scheduled injections taken per participant | 12 months
  The percentage of scheduled injections taken per participant is calculated as the proportion of actual number of injections with Ngenla or daily growth hormone used from the total number of expected injections.
Change from baseline in Life Interference Questionnaire-Growth Hormone Deficiency I (LIQ-GHD I) questionnaire | 12 months
  The LIQ-GHD I instrument uses either a 5 point scale from never to always or very easy to very difficult or a 7 point scale from extremely convenient to extremely inconvenient.
  It contains the following subscales:
  * Pen ease of use
  * Ease of the injection schedule
  * Satisfaction with overall treatment experience
  * Willingness to continue injection schedule
  * Patient life interference
  * Number of missed injections during the past 4 weeks(two questions asking for number of missed injections and reasons)
  * Caregiver life interference
Change from baseline in Quality of Life in Short Stature Youth (QoLISSY) questionnaire for patients and for caregivers | 12 months
  The QoLISSY questionnaire is a 5 point scale from not at all/never to extremely/always.
  It evaluates the following health related quality of life domains for participants and their caregivers:
  * Physical impact of height
  * Social impact of height
  * Emotional impact of height
Healthcare practitioner (HCP) preference survey | 12 months
  HCP preference and satisfaction survey for treatment regimen and treatment experience (daily or weekly injections or no preference) and satisfaction rated from very satisfied to very dissatisfied.
Change from baseline in effectiveness evaluations for Ngenla and daily growth hormone | 12 month
  Height in cm, weight in kg, and BMI in kg/m2 at diagnosis and follow-up visits and annualized height velocity in cm.
Presence or absence of factors influencing adherence | 12 months
  Lifestyle factors are assessed:
  * travel, illness, overnight sleep
  * injection administration by caregiver/nurse or self-administration Number of concomitant medications and route of administration are collected
Mean Adherence To Ngenla and daily growth hormone for age subgroups. | 12 months
  -Different age groups: 3-7 years/8-11 years/12-16 years The adherence for Ngenla and daily growth hormone follows the medication possession ratio definition(MPR). The MPR is calculated from the total number of injections used and collected in the Smart Sharps Bin™ .
Mean Adherence To Ngenla and daily growth hormone for switch participants | 12 months
  - Switch participants: dGH to Ngenla and vice versa The adherence for Ngenla and daily growth hormone follows the medication possession ratio definition(MPR). The MPR is calculated from the total number of injections used and collected in the Smart Sharps Bin™ .
Mean Adherence To Ngenla and daily growth hormone for naive/non-naive subgroups. | 12 months
  - Treatment naïve vs non-naïve (either dGH or Ngenla) The adherence for Ngenla and daily growth hormone follows the medication possession ratio definition(MPR). The MPR is calculated from the total number of injections used and collected in the Smart Sharps Bin™ .
Number of participants who discontinued Ngenla or daily growth hormone | 12 months
  Persistency/discontinuation is evaluated at specific time windows, after patients stop utilizing the sharps bin.
Percent of participants who discontinued Ngenla or daily growth hormone | 12 months
  Persistency/discontinuation is evaluated at specific time windows, after patients stop utilizing the sharps bin.
Number of participants who switch growth hormone treatment | 12 months
  Number of participants who switch from daily to weekly GH injections or from weekly to daily GH injections is reported.
Percentage of participants who switch growth hormone treatment | 12 months
  Percentage of participants who switch from daily to weekly GH injections or from weekly to daily GH injections is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0311024